CLINICAL TRIAL: NCT02452606
Title: Clock and Narcolepsy Genetic Variants and the Effects of Stalevo® (Levodopa/Carbidopa/Entacapone) on Sleep Disorders in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sun Ju Chung, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0241
Record Dates: First submitted 2015-05-14; First posted 2015-05-22 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Parkinson Disease; Sleep Disorders
Keywords: Stalevo; sleep disturbance; central circadian clock; narcolepsy
MeSH Terms: conditions — Parkinson Disease; Sleep Wake Disorders; Parasomnias; Narcolepsy | interventions — Stalevo; Levodopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stalevo® (Experimental): Participants who are assigned to Stalevo Arm will take Stalevo® at bedtime for 3 month.
  Interventions: Drug: Stalevo®

INTERVENTIONS:
Drug: Stalevo® — * Sleep disorders in Parkinson's disease
  * Analysis by Parkinson's Disease Sleep Scale(PDSS) scores.
  * If the PDSS score is improving at least 15 percent than the baseline score, It can be determined to be effective.
  Other Names: Levodopa/Carbidopa/Entacapone

SUMMARY:
The purpose of this study is to investigate the genetic variants of clock and narcolepsy genes that determine the therapeutic effects of Stalevo® on the quality of sleep in patients with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with PD in accordance with UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria (Hughes AJ, et al. 1992).
2. Patients with PD who have wearing off phenomenon.
3. Patients with PD with Hoehn and Yahr stage 1-4.
4. Patients with PD who have sleep problems (PDSS score ≤120 or Epworth Sleepiness Scale(ESS) score ≥ 8).
5. Patients with PD who showed Montreal Cognitive Assessment (MoCA) score ≥15.
6. Patients with PD who have no major depression (Geriatric depression scale, GDS ≤ 24)

Exclusion Criteria:

1. Secondary parkinsonism
2. Parkinson-plus syndromes (multiple system atrophy, progressive supranuclear palsy, and corticobasal degeneration.
3. Patients with PD who have history of severe side effect of Stalevo®.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The correlation of the genetic variants of central circadian clock and narcolepsy genes with regard to the treatment effect of Stalevo® in sleep disturbance of parkinson's disease. | 2 years
  To determine whether the genetic variants of clock and narcolepsy genes are associated with the effectiveness of Stalevo® in bedtime on the quality of sleep in PD patients with motor fluctuation.

SECONDARY OUTCOMES:
The effectiveness of Stalevo® in bedtime on the quality of sleep in PD patients with motor fluctuation (using Parkinson's Disease Sleep Scale) | up to 3 months from enrollment.
  To determine whether Stalevo® in bedtime improves the quality of sleep in PD patients with motor fluctuation using Parkinson's Disease Sleep Scale.
The effectiveness about improving the EDS(Excessive daytime sleepiness) in PD patients with motor fluctuation after taking Stalevo® in bedtime. | up to 3 months from enrollment.
  Excessive daytime sleepiness (EDS) is characterized by persistent sleepiness and often a general lack of energy, even after apparently adequate or even prolonged night time sleep. EDS can be considered as one of features of sleep disturbance in parkinson's disease. It will be assessed using a composite measurement consisting of Unified Parkinson's Disease Rating Scale (UPDRS), Hoehn and Yahr stage, Parkinson's Disease Sleep Scale (PDSS), Epworth Sleepiness Scale (ESS), Parkinson's Disease Wearing Off Questionnaire-9 (PDWOQ-9), and Parkinson's Disease Quality of Life Questionnaire-39 (PDQ-39).
The effectiveness about improving the morning motor symptoms in PD patients with motor fluctuation after taking Stalevo® in bedtime. | up to 3 months from enrollment
  To determine whether Stalevo® in bedtime improves the morning motor symptoms in PD patients with motor fluctuation. It will be assessed using a composite measurement consisting of Unified Parkinson's Disease Rating Scale (UPDRS), Hoehn and Yahr stage, Parkinson's Disease Sleep Scale (PDSS), Epworth Sleepiness Scale (ESS), Parkinson's Disease Wearing Off Questionnaire-9 (PDWOQ-9), and Parkinson's Disease Quality of Life Questionnaire-39 (PDQ-39).

CONTACTS AND LOCATIONS:
Overall Officials: Sun Ju Chung, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea